CLINICAL TRIAL: NCT02217774
Title: MGUIDE MORE Dental Implant Planning System- Clinical Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: MIS Implant Technologies, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0210-14-RMB CTIL; 0210-14-RMB (Other: Rambam Health Care Campus Internal Review Board)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Focus of Study: Computer-Aided Design/Instrumentation
Keywords: Computer-Aided Design/instrumentation; Cone-Beam Computed Tomography; Dental Implant; MGuide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MGUIDE assisted implant placement (Experimental): Implant placement, using MGUIDE MORE system for implant planning and placement
  Interventions: Device: MGUIDE MORE

INTERVENTIONS:
Device: MGUIDE MORE — MGUIDE MORE System (MGS), consisting of MGUIDE MORE software, MGUIDE MORE surgical kit and MGUIDE MORE template, will be used for planning, drilling and inserting dental implants.

SUMMARY:
The aim of the present study is to assess the accuracy of MGUIDE MORE System (MGS), consisting of MGUIDE MORE software, MGUIDE MORE surgical kit and MGUIDE MORE template by evaluating the difference between planned and actual implant positions on pre- and post-operative CBCTs.

DETAILED DESCRIPTION:
Patients, attending the Department of Periodontology at the Rambam School of Graduate Dentistry, who are scheduled for implant therapy, will be screened for the study. Patients will be referred for CBCT of the upper/lower jaw as appropriate. DICOM data of the patient will be uploaded to MGUIDE software and used for diagnosis and treatment planning of the case. Surgery will be performed using MGUIDE MORE template and MGUIDE MORE surgical kit. Pre-operative and post-operative CBCT will be used for assessment of the difference between planned and actual implant positions.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated inform consent form.
* Age between 18+.
* Patient expresses his wish to restore the missing tooth/teeth with dental implants.
* Patient is examined and found suitable for implant therapy
* Patient can open mouth sufficiently for preparation and placement of dental implants using the contra-angle handpiece and drills.
* CBCT is required for proper diagnosis and treatment planning.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08-23 (Actual); Study Completion 2015-08-23 (Actual)

PRIMARY OUTCOMES:
Deviation from planning | 0-14 days after implant placement
  To assess shoulder and apex deviations in milimeters between planned and actual implant position and to assess angular deviation in degrees, of actual implant position vs. planned implant position

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Horwitz, DMD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] Horwitz J, Zuabi O, Machtei EE. Accuracy of a computerized tomography-guided template-assisted implant placement system: an in vitro study. Clin Oral Implants Res. 2009 Oct;20(10):1156-62. doi: 10.1111/j.1600-0501.2009.01748.x. Epub 2009 Jun 10. PMID 19519787